CLINICAL TRIAL: NCT04031144
Title: Effect of Ultrafiltration Before Weaning From Cardiopulmonary Bypass on Post-bypass Coagulation Function in Cardiac Surgery
Brief Title: Ultrafiltration on Coagulation Function in Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Konkuk University Medical Center (Other)
Responsible Party: Principal Investigator, Tae-Yop Kim, MD PhD, Professor of Anesthesiology, Konkuk University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KUMC 2019-05-008
Record Dates: First submitted 2019-07-21; First posted 2019-07-24 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Cardiac Valve Disease
Keywords: coagulation; ultrafiltration; cardiac surgery
MeSH Terms: conditions — Heart Valve Diseases; Thrombosis | interventions — Ultrafiltration

STUDY DESIGN:
Intervention Model Description: Patients with reduced clot strength before applying ultrafiltration (patients with MCF in ROTEM-EXTEM less than the cut-off value, determined by preliminary analyses, n=30).
  ROC analysis of the preliminary data was performed, and the cut-off value was 50.5 mm.
  The sample size of the present study is determined by using these data. The minimum sample size to detect the observed difference after applying ultrafiltration was 26. Considering 50% possible loss, 39 patients will be recruited for the primary analysis.
  Patients scheduled for elective cardiac surgery with cardiopulmonary bypass are recruited first, and the data from patients with MCF <50.5 mm will be included in the final analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ultrafiltration (Experimental): Ultrafiltration is applied at the end of cardiopulmonary bypass. Maximal clot formation (MCF) of ROTEM-EXTEM tracing is reduced before applying the ultrafiltration.
  Interventions: Procedure: Ultrafiltration

INTERVENTIONS:
Procedure: Ultrafiltration — At the end of CPB procedure, free water is partly removed by ultrafiltration to increase relative mass of red blood cell and plasma components.

SUMMARY:
To determine the effect of modified ultrafiltration, which is usually employed for reducing free water at the end of cardiopulmonary bypass (CPB), on coagulation profile in patients undergoing cardiac surgery

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing elective cardiac surgery with cardiopulmonary bypass (CPB)
* maximal clot formation (MCF) in ROTEM-EXTEM is reduced (< 50.5 mm before applying ultrafiltration)

Exclusion Criteria:

* transfusion of packed RBC> 3 units during CPB
* total ultrafiltration volume < 250 ml
* hyperfibrinolysis (lysis% > 10%) before applying ultrafiltration

Ages: 19 Months to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2020-01-30 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Change of Maximal clot formation (MCF) in rotational thromboelastometry, EXTEM assay | 5 min-before and 5 min-after applying ultrafiltration
  change of MCF in EXTEM assay before and after applying ultrafiltration

SECONDARY OUTCOMES:
Change of Clotting time (CT) in rotational thromboelastometry, EXTEM assay | 5 min-before and 5 min-after applying ultrafiltration
  change of CT in EXTEM assay before and after applying ultrafiltration
Change of Maximal clot formation at 5 min (A5) in rotational thromboelastometry, FIBTEM assay | 5 min-before and 5 min-after applying ultrafiltration
  change of A5 in FIBTEM assay before and after applying ultrafiltration
Change of Percent of lysis (lysis%) in rotational thromboelastometry, EXTEM assay | 5 min-before and 5 min-after applying ultrafiltration
  change of lysis% before and after applying ultrafiltration
Hematocrit (Hct) change | 5 min-before and 5 min-after applying ultrafiltration
  change of Hct before and after applying ultrafiltration

CONTACTS AND LOCATIONS:
Locations (1):
- Konkuk University Medical Center, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided